CLINICAL TRIAL: NCT02650466
Title: Nanopulse Efficacy Study for the Treatment of Common Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Stefani Takahashi, Associate Professor, Director, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EnI-13129
Record Dates: First submitted 2015-11-12; First posted 2016-01-08 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Common Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nanopulse treatment (Experimental): The study will be a single center, open label, non-randomized clinical trial that will provide efficacy data for the treatment of common warts by the Nanopulse system in terms of efficacy and cosmetic outcome with 1 - 4 application (treatment) sessions. All subjects will receive a minimum number of applications per discrete skin wart lesion. Up to 4 warts per subject will be treated with the Nanopulse device. The wart will be debulked to the point of pinpoint bleeding prior to the initial application. The subject will return after 1 week for an evaluation visit and at 4 weeks for a second treatment and 2 additional monthly treatments if warranted. If the subject is declared clinically clear at any of the application visits, they will be placed into follow up. The minimum number of treatments per wart is one and the maximum is 4. They will return at the 12 week point post last visit for final assessment and evaluation.
  Interventions: Device: Nanopulse System

INTERVENTIONS:
Device: Nanopulse System — The Nanopulse System consists of an electrical pulse generator, a handpiece, and a detachable applicator tip at the end of the handpiece that interfaces with the treatment area on the skin. The detachable applicator tip delivers the pulses to the skin through five 3 mm long needle electrodes (27 gauge). The applied electric field, is limited to the space enclosed by the 4 outer electrodes in the applicator tip. An inert, water based gel is applied to the skin and the applicator tip before making contact between subject and applicator tip to ensure that there are no air gaps present between the electrodes through which electrical arcing could occur while pulses are being delivered to the subject. The Applicator Tips are designed for single patient use, and are sterilized prior to first use and between treatment sessions using a standard steam autoclave.

SUMMARY:
The purpose of this study is to determine if the Nanopulse System can be used to clear common wart lesions on the skin. The Nanopulse System uses a series of low energy, high voltage pulses, each one several billionths of a second in duration, to effectively kill the target tissue contained within the applicator tip electrodes with minimal damage to surrounding tissue. Efficacy and patient outcomes are expected to equal or surpass current treatment modalities in terms of increased ease of use, faster patient healing and minimal scarring with fewer complications resulting from treatment.

The device emits significantly less energy than existing electro-surgery or electro-cautery equipment and is believed to be similar to laser therapy treatment of warts. Trained clinicians can usually diagnose warts based by their appearance and location . Non-genital warts are subcategorized into common, periungual, flat, filiform, and plantar types. Common warts are benign, often skin-colored, or brown-grey, rough, bumpy growths on the hands and feet (caused by Human Papilloma Virus type 2) . Common warts in individuals without any immune deficiencies are low risk and are the focus of this study.Based upon the preclinical profile of the Nanopulse device, particularly its safety profile and its effect on transformed cells, it is hypothesized that application of pulses from the Nanopulse System , will result in complete clinical clearance of Common Wart lesions with minimal scarring.

DETAILED DESCRIPTION:
Study Objective: The objective of this study is to indicate whether the Nanopulse System is efficacious for use in clearing common warts.

The primary objective of this study is to gather lesion clearance data on common warts after application of pulses from the Nanopulse System and determine the optimal number of treatments necessary. Clearance will be measured by clinical observation.

Other objectives of the study include gathering efficacy data on the use of the Nanopulse System for treating common warts in terms of:

1.) Safety in a clinical setting in terms of minimal adverse events over the course of the trial; 2.) Cosmetic results during the healing process and cosmetic outcome; 3.)Effects of 1, 2, 3 or 4 treatments in terms of clearance and cosmetic outcome for each treated wart; 4.)Subject impressions immediately following application of pulses; 5.)Subject satisfaction with the treatment and cosmetic outcome during and following the healing process; 6) Device performance and clinical feedback under actual clinical conditions and to gather information on design features that may be modified to optimize the device.

ELIGIBILITY:
Inclusion Criteria:

* Only Common Warts will be included as study lesions.
* Only discrete common warts in a single 5cm x 5cm anatomical area can be included as study lesions. Up to 4 discrete common warts that meet this criteria can be treated per subject. The 5cm x 5cm area must not have more than 2 warts present at the time of screening and warts outside each area must be at least 2cm away from warts included as study lesions. Please Note: A single digit (e.g. finger) can represent a 5cm x 5cm area, and a lesion within the area can be included as a study lesion UNLESS it is on the inside surface of a digit where there are wart lesions present on the surface of an adjacent digit that would be within 1 cm of touching the potential study lesion when the surfaces of the digits are in contact with one another.
* Subject's lesion may have been treated with over-the-counter treatments, but not by any prescription medicine, surgery, or destructive procedure (i.e., cryotherapy) within four weeks of the date the subject is recruited into the study.
* Subject's wart and the subject must be suitable candidates for usual Standard of Care treatments. Standard of care for common warts is defined as curettage and electrodesication, cryotherapy, topical therapy or surgery.
* Subject must be competent to provide informed consent.
* If the subject is female, and of childbearing potential, subject must be actively practicing a clinically acceptable form of birth control.
* Subject's medical evaluation during their screening visit does not indicate any findings of clinical significance relevant to participating in study.
* Subject has been informed of their options for standard of care for the lesion type outside of the study.

Exclusion Criteria:

* Subjects not meeting all inclusion criteria should be excluded.
* Subjects who have lesions within the 5cm x 5cm anatomical area under study which are painful or have been noticeably changing just prior to the time of screening.
* Periungual warts are excluded from the study as study lesions. Subject is to be informed that these warts will not be treated during the duration of the study.
* Lesions on the face are excluded from the study as study lesions.
* Lesions which are diagnosed as flat warts, filiform warts, plantar warts, and genital warts are excluded from the study as study lesions. Subject is to be informed that these warts will not be treated during the duration of the study.
* Subjects who are using or intend to use any other warts therapy concomitantly during the study period or within 4 weeks of their screening visit.
* Subjects who are not capable of undergoing surgical standard of care treatment for common warts due to mental or physical limitations.
* Subjects in whom a minor surgical procedure is contraindicated (e.g. under advice of their own caring clinician).
* Subjects who have an implanted artificial heart valve or other prosthesis requiring prophylactic antibiotic coverage for minor surgical procedures.
* Subjects who have an implanted cardiac pacer or defibrillator or other similar life sustaining implanted electrical device.
* Subjects who have had any cosmetic or therapeutic procedure (e.g. use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within 2cm of targeted area and margins within 4 weeks of the screening visit and within 10cm of treatment area during the study.
* Subjects who are immunosuppressed either due to an existing medical diagnosis, or are currently using medications that suppress the immune system (e.g. cyclosporine, prednisone, methotrexate, alefacept, infliximab) or have used these medications within 8 weeks of the screening visit or anytime during the study.
* Topical immunomodulators (imiquimod, steroid creams) within 4 weeks of the screening visit or any time during the study.
* Prolonged or excessive exposure to ultra-violet light within 2 weeks prior to screening visit or any time during the study.
* Subjects who, if female, know that they are currently pregnant or are lactating and actively breastfeeding.
* Under the Investigator's authority to exclude any participant at his/her discretion, participation in this study is not recommended for this Subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2016-08-20 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefani Takahashi, MD, Principal Investigator — University of Southern California
Locations (1):
- Huntington Medical Foundation, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nanopulse Treatment: The study will be a single center, open label, non-randomized clinical trial that will provide efficacy data for the treatment of common warts by the Nanopulse system in terms of efficacy and cosmetic outcome with 1 - 4 application (treatment) sessions. All subjects will receive a minimum number of applications (n=1 application) per discrete skin wart lesion. Up to 4 warts per subject will be treated with the Nanopulse device. The wart will be debulked to the point of pinpoint bleeding prior to the initial application. The subject will return after 1 week for an evaluation visit and at 4 weeks for a second treatment and 2 additional monthly treatments if warranted. If the subject is declared clinically clear at any of the application visits, they will be placed into follow up. They will return at the 12 week point post last visit for final assessment and evaluation.
  Nanopulse System: The Nanopulse System consists of an electrical
Period: Overall Study
Arm/Group | Nanopulse Treatment
Started | 24
Completed | 17
Not Completed | 7
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: number of warts treated
Groups:
- Nanopulse Treatment: The Nanopulse System consists of an electrical pulse generator, a handpiece, and a detachable applicator tip at the end of the handpiece that interfaces with the treatment area on the skin. The applicator tip delivers pulses to the skin through needle electrodes. The Applicator Tips are designed for single patient use, and are sterilized prior to first use and between treatment sessions using a standard steam autoclave.
  All subjects will receive a minimum number of applications per discrete skin wart lesion (n=1 application). Up to 4 warts per subject will be treated. The wart will be debulked prior to the initial application. The subject will return after 1 week for an evaluation visit, at 4 weeks for a second treatment and up to 2 additional monthly treatments. Subjects will be evaluated at each application visit and placed in follow-up when they are declared clinically clear. They will return at the 12 week point post last visit for final assessment and evaluation.
Arm/Group | Nanopulse Treatment
Number analyzed (Participants) | 24
Number analyzed (number of warts treated) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian (non-Hispanic) | 13
  Hispanic Latino | 2
  African-American | 1
  Asian/SE Islan | 7
  Native American | 0
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Clinical Clearance of Warts
Description: Response rate is defined in each case in terms of no effect (NE=2), partial response (PR=1), or complete response (CR=0). No Effect (NE) would indicate no clinically apparent reduction in lesion size, Partial Response (PR) would indicate a reduction in lesion size, and Complete Response (CR) would indicate no evidence of the lesion detected.
Time Frame: 168 days after first treatment application
Population: The total number of participants who completed the study equals 17. But because one participant had 3 warts that received treated with differing results, they are counted twice (for that participant, one wart cleared and two showed no effect).
Measure: Number; unit: # of warts
Units Other Than Participants: # of warts treated
Groups:
- Partially Removed(1): wart size has been reduced in height and width during treatment.
Arm/Group | Partially Removed(1)
Number analyzed (Participants) | 17
Number analyzed (# of warts treated) | 19
# of warts
  Cleared | 13
  Partially Removed | 4
  No Effect | 2

2. Secondary Outcome: Total Number of Adverse Events That Occur During the Course of the Study
Description: Number of participants who experience an adverse event, regardless of whether they completed the study, will be aggregated through study completion. Both anticipated and unanticipated adverse events will be reported.
Time Frame: an average of 140 days
Population: During initial treatment of a wart on a digit, mild pain radiated up the finger from the wart at time of treatment. The pain persisted for 30min. P.O. Tylenol was provided at the time treatment. This did not re-occur during treatments 2,3 and 4.
Measure: Number; unit: participants
Units Other Than Participants: # of warts treated
Groups:
- Number of Adverse Events: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
  For those anticipated adverse reactions which are not present before the first application procedure and are rated at a severity level above minimal or mild will be recorded at the time of occurrence. The adverse event will be reported to the sponsor, and will be followed by study personnel through to its resolution. All unanticipated adverse reactions, regardless of their severity, will be recorded as adverse events and reported to the sponsor.
Arm/Group | Number of Adverse Events
Number analyzed (Participants) | 24
Number analyzed (# of warts treated) | 30
participants | 1

3. Secondary Outcome: Total Number of Serious Adverse Events That Occur During the Course of the Study
Description: Number of participants, regardless of whether they completed the study, who experience serious adverse events will be aggregated through study completion from the clinical report forms and reported at the end of the study.
Time Frame: an average of 140 days
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Serious Adverse Events
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data (including serious adverse event data) from 24 participants was collected on average for: 209 days (Range: 168-300 days) for the 17 participants who completed the study; and, 79 days (Range:0-217 days) from the 7 participants who did not complete the study.
Description: For each adverse event, the details of and circumstances will be recorded at the site and evaluated by the investigator in terms of relatedness, seriousness and the degree to which the event was anticipated.The adverse event will be reported to the sponsor and the Institutional Review Board; and will be followed by study personnel through to its resolution. All unanticipated adverse reactions, regardless of their severity, will be recorded as adverse events and reported to the sponsor.
Arm/Group | Nanopulse Treatment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nanopulse Treatment (N=24)
Local Sensory Abnormality (Skin and subcutaneous tissue disorders) | 1 (1) — During initial treatment of a wart on a digit, mild pain radiated up the finger from the wart at time of treatment. The pain persisted for 30min.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No